CLINICAL TRIAL: NCT01175850
Title: Randomized Trial of IN.PACT Admiral(TM) Drug Coated Balloon vs Standard PTA for the Treatment of SFA and Proximal Popliteal Arterial Disease
Brief Title: Randomized Trial of IN.PACT Admiral® Drug Coated Balloon vs Standard PTA for the Treatment of SFA and Proximal Popliteal Arterial Disease
Acronym: INPACT SFA I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P990
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug-Coated Balloon (DCB) (Experimental): IN.PACT Admiral: Balloon Angioplasty
  Interventions: Device: Drug-Coated Balloon (DCB)
- Standard PTA (Active Comparator): Standard Percutaneous Transluminal Angioplasty (PTA) Balloon: Balloon Angioplasty
  Interventions: Device: PTA Balloon: Balloon Angioplasty

INTERVENTIONS:
Device: Drug-Coated Balloon (DCB) — balloon dilatation and provisional stenting with IN.PACT DCB
  Arms: Drug-Coated Balloon (DCB)
Device: PTA Balloon: Balloon Angioplasty — balloon dilatation and provisional stenting with standard non-coated PTA balloon
  Arms: Standard PTA

SUMMARY:
The objective of this Study is to evaluate the safety and efficacy of the IN.PACT Admiral® drug coated PTA balloon, utilized for the dilatation of the narrowed sections of the artery, as compared to other standard (non drug coated) PTA balloons. The IN.PACT Admiral, besides the mechanical dilatation effect typical of all PTA balloons, releases a drug (paclitaxel) from the balloon surface into the vessel walls. This drug absorption is intended to limit the chances and the entity of artery re-narrowing over time.

DETAILED DESCRIPTION:
The efficacy of the IN.PACT Admiral balloon will be evaluated by assessing the primary patency rate of the treated arteries in the thighs of all patients included in the Study. Primary patency is a measure of the durability up to 1 year of the free lumen in the artery as restored during the procedure and is based on:

* the need for re-dilatation of the previously treated vessel segment
* an ultrasound examination The safety of the IN.PACT Admiral will be assessed by evaluating the incidence of deaths, amputations and re-dilatation of the pre-treated arteries in all patients included in the Study.

The IN.PACT SFA Trial enrolled in 2 phases: IN.PACT SFA I and IN.PACT SFA II. The 150-patient IN.PACT SFA I phase is intended to support the second phase IN.PACT SFA II IDE trial with congruent design and protocol. Aggregate data from the two phases is intended to provide statistical power for the 12-month primary safety and effectiveness endpoints.

ELIGIBILITY:
General Inclusion Criteria:

* Age ≥18 years and ≤85 years
* Patient or patient's legal representative is informed of the nature of the study, agrees to participate and has signed an EC approved consent form

Angiographic Inclusion Criteria:

- Target vessel is the superficial femoral artery and/or proximal popliteal artery (above the knee)

General Exclusion Criteria:

* Patient unwilling or unlikely to comply with follow-up schedule
* Stroke or STEMI within 3 months prior enrolment

Angiographic Exclusion Criteria:

- Acute or sub-acute thrombus in the target vessel

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, Prof Dr. Med, Principal Investigator — Klinikum Rosenheim
Locations (1):
- Klinikum Rosenheim Institut für Diagnostische und Interventionelle Radiologie, Rosenheim, Pettenkoferstr, Germany

REFERENCES:
- [Derived] Krishnan P, Farhan S, Schneider P, Kamran H, Iida O, Brodmann M, Micari A, Sachar R, Urasawa K, Scheinert D, Ando K, Tarricone A, Doros G, Tepe G, Yokoi H, Laird J, Zeller T. Determinants of Drug-Coated Balloon Failure in Patients Undergoing Femoropopliteal Arterial Intervention. J Am Coll Cardiol. 2022 Sep 27;80(13):1241-1250. doi: 10.1016/j.jacc.2022.06.043. PMID 36137674
- [Derived] Shishehbor MH, Schneider PA, Zeller T, Razavi MK, Laird JR, Wang H, Tieche C, Parikh SA, Iida O, Jaff MR. Total IN.PACT drug-coated balloon initiative reporting pooled imaging and propensity-matched cohorts. J Vasc Surg. 2019 Oct;70(4):1177-1191.e9. doi: 10.1016/j.jvs.2019.02.030. PMID 31543165
- [Derived] Laird JA, Schneider PA, Jaff MR, Brodmann M, Zeller T, Metzger DC, Krishnan P, Scheinert D, Micari A, Wang H, Masters M, Tepe G. Long-Term Clinical Effectiveness of a Drug-Coated Balloon for the Treatment of Femoropopliteal Lesions. Circ Cardiovasc Interv. 2019 Jun;12(6):e007702. doi: 10.1161/CIRCINTERVENTIONS.118.007702. Epub 2019 Jun 14. PMID 31195825
- [Derived] Schneider PA, Laird JR, Doros G, Gao Q, Ansel G, Brodmann M, Micari A, Shishehbor MH, Tepe G, Zeller T. Mortality Not Correlated With Paclitaxel Exposure: An Independent Patient-Level Meta-Analysis of a Drug-Coated Balloon. J Am Coll Cardiol. 2019 May 28;73(20):2550-2563. doi: 10.1016/j.jacc.2019.01.013. Epub 2019 Jan 25. PMID 30690141
- [Derived] Schneider PA, Laird JR, Tepe G, Brodmann M, Zeller T, Scheinert D, Metzger C, Micari A, Sachar R, Jaff MR, Wang H, Hasenbank MS, Krishnan P; IN.PACT SFA Trial Investigators. Treatment Effect of Drug-Coated Balloons Is Durable to 3 Years in the Femoropopliteal Arteries: Long-Term Results of the IN.PACT SFA Randomized Trial. Circ Cardiovasc Interv. 2018 Jan;11(1):e005891. doi: 10.1161/CIRCINTERVENTIONS.117.005891. PMID 29326153
- [Derived] Tepe G, Laird J, Schneider P, Brodmann M, Krishnan P, Micari A, Metzger C, Scheinert D, Zeller T, Cohen DJ, Snead DB, Alexander B, Landini M, Jaff MR; IN.PACT SFA Trial Investigators. Drug-coated balloon versus standard percutaneous transluminal angioplasty for the treatment of superficial femoral and popliteal peripheral artery disease: 12-month results from the IN.PACT SFA randomized trial. Circulation. 2015 Feb 3;131(5):495-502. doi: 10.1161/CIRCULATIONAHA.114.011004. Epub 2014 Dec 3. PMID 25472980

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The IN.PACT SFA Trial was designed as a two-phase randomized trial. IN.PACT SFA I, the first phase was conducted in Europe with 150 subjects enrolled. IN.PACT SFA II, the second phase, was conducted in the US with 181 subjects enrolled. The data from both phases of the IN.PACT SFA Trial have been pooled and comprise the pivotal trial data.
Groups:
- Drug-Coated Balloon (DCB): Paclitaxel drug-coated angioplasty balloon
  IN.PACT Admiral Drug-Coated Balloon: Subjects will be randomized 2:1 to the IN.PACT Admiral Drug-Coated Balloon Arm or to the standard angioplasty balloon Arm
- Standard PTA: Standard angioplasty balloon without Paclitaxel drug-coating
  Standard angioplasty balloon: Subjects will be randomized 2:1 to the IN.PACT Admiral Drug-Coated Balloon Arm or to the standard angioplasty balloon Arm
Period: IN.PACT SFA I Phase
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Started | 99 | 51
Completed | 88 | 49
Not Completed | 11 | 2
Period: IN.PACT SFA II Phase
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Started | 121 | 60
Completed | 109 | 55
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA | Total
Number analyzed (Participants) | 220 | 111 | 331
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (9.5) | 68.0 (9.2) | 67.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 36 | 113
  Male | 143 | 75 | 218

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency
Description: Primary patency is defined as freedom from clinically-driven target lesion revascularization (TLR) or restenosis as determined by duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) ≤ 2.4.
Time Frame: 12 Month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 191 | 103
Percentage of participants | 82.2 | 52.4
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p < 0.001, Z-test; Z-test of two proportions was used to compare treatment groups for all randomized subjects

2. Primary Outcome: Primary Safety Composite
Description: Primary safety composite is defined as freedom from death through 30 days or target limb major amputation or clinically-driven target vessel revascularization (CD-TVR) within 12 months post index procedure.
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of Participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 207 | 107
Percentage of Participants | 95.7 | 76.6
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Secondary Outcome: Major Adverse Events (MAE) Composite
Description: Major Adverse Events (MAE) composite defined as all-cause death, clinically-driven target vessel revascularization (CD-TVR), major target limb amputation, thrombosis at the target lesion site
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 207 | 107
Percentage of participants | 6.3 | 24.3
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Secondary Outcome: All-cause Death
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 207 | 107
percentage of participants | 1.9 | 0.0
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.926, Chi-squared

5. Secondary Outcome: Target Vessel Revascularization (TVR)
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 207 | 107
Percentage of participants | 4.8 | 23.4
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p < 0.001, Chi-squared

6. Secondary Outcome: Target Lesion Revascularization (TLR)
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 207 | 107
Percentage of participants | 2.9 | 20.6
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p < 0.001, Chi-squared

7. Secondary Outcome: Time to First Clinically Driven Target Lesion Revascularization (CD-TLR)
Description: Clinically-driven target lesion revascularization (CD-TLR) is defined as any re-intervention within the target lesion due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure baseline.
Time Frame: 12 month
Population: Includes all subjects who experienced a CD-TLR.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 5 | 22
Days | 144.6 (159.6) | 201.9 (90.9)
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.859, Chi-squared

8. Secondary Outcome: Major Target Limb Amputation
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: percentage of amputations
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 207 | 107
percentage of amputations | 0 | 0
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p > 0.999, Chi-squared

9. Secondary Outcome: Thrombosis at the Target Lesion
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 207 | 107
Percentage of participants | 1.4 | 3.7
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.096, Chi-squared

10. Secondary Outcome: Primary Sustained Clinical Improvement
Description: Freedom from target limb amputation, target vessel revascularization (TVR), and increase in Rutherford class. Rutherford classification is a clinical staging system that is used to describe peripheral arterial disease.
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: percentage of particpants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 196 | 106
percentage of particpants | 85.2 | 68.9
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p < 0.001, Chi-squared

11. Secondary Outcome: Secondary Sustained Clinical Improvement
Description: Freedom from target limb amputation and increase in Rutherford class.
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 196 | 104
percentage of participants | 89.3 | 84.6
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.121, Chi-squared

12. Secondary Outcome: Duplex-defined Binary Restenosis (Peak Systolic Velocity Ratio (PSVR) >2.4).
Description: Duplex ultrasound measurement that measures the peak systolic velocity of blood (cm/sec) within a lesion divided by the peak velocity of blood (cm/sec) proximal to the lesion.
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 188 | 86
Percentage of participants | 16.5 | 33.7
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.001, Chi-squared

13. Secondary Outcome: Duplex-defined Binary Restenosis (Peak Systolic Velocity Ratio >3.4).
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Number; unit: Percentage of particpants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 178 | 84
Percentage of particpants | 7.3 | 21.4
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p < 0.001, Chi-squared

14. Secondary Outcome: Change From Baseline in Quality of Life Assessment by EuroQol Group 5-Dimension Self Report Questionnaire (EQ5D) at Month 12
Description: Quality of life assessment by EQ5D at 1 year compared to baseline. EQ5D is a standardised measure of health status and economic appraisal. The EQ5D consists of the EQ5D descriptive system which comprises the following variables for the 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: (1) no problems, (2) some problems, (3) extreme problems. A complex algorithm that took individual dimensions and generated an overall score was used.
  EQ5D health state is used in the algorithm to calculate an overall score where - 0.109 = 'worst possible outcome' and 1.000 = 'best possible outcome'.
Time Frame: Baseline to 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 193 | 102
Units on a scale | 0.1059 (0.2089) | 0.0730 (0.1951)
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.095, Chi-squared

15. Secondary Outcome: Change From Baseline in Walking Capacity Assessment by Walking Impairment Questionnaire (WIQ) at 12 Months
Description: Walking capacity assessment by WIQ at 1 year compared to baseline. WIQ is a quality of life questionnaire that was specifically designed to assess the degree of impairment experienced by patients with claudication.
  Clinical outcomes were assessed by patients responses to question 1A. Question 1A is specific for calf or buttocks claudication and is used to create a summary score for analysis. Question 1A is expressed on a scale of 0% (unable to perform because of severe claudication) to 100% (no impairment).
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 196 | 104
Units on a scale | 72.7 (31.4) | 73.6 (29.5)
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.590, Chi-squared

16. Secondary Outcome: Device Success
Description: Device success is defined as successful delivery, balloon inflation and deflation and retrieval of the intact study device without burst below rated burst pressure (RBP).
Time Frame: Day 1
Population: Total number of devices used in the ITT population (n=331).
Measure: Number; unit: Percentage of devices
Units Other Than Participants: Devices
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 220 | 111
Number analyzed (Devices) | 311 | 130
Percentage of devices | 99.0 | 98.5
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.302, Chi-squared

17. Secondary Outcome: Procedural Success
Description: Procedural success is defined as obtainment of ≤30% residual stenosis by visual estimate (with or without stenting)
Time Frame: Day 1
Population: Intention-to-Treat (ITT) (n=331)
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 220 | 111
Percentage of participants | 99.5 | 98.2
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.111, Chi-squared

18. Secondary Outcome: Clinical Success
Description: Clinical success is defined as procedural success without procedural complications (death, stroke, major target limb amputation, thrombosis of the target lesion, or target vessel revascularization (TVR)) prior to discharge.
Time Frame: Day 1
Population: Intention-to-Treat (ITT) (n=331)
Measure: Number; unit: Percentage of participants
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 220 | 111
Percentage of participants | 99.1 | 97.3
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.103, Chi-squared

19. Secondary Outcome: Days of Hospitalization Due to the Index Lesion
Description: Days of hospitalization from procedure through 12 month.
Time Frame: 12 month
Population: Intention-to-Treat (ITT) (n=331) that excludes subjects who did not have evaluable data at the reporting timeframe.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Number analyzed (Participants) | 219 | 111
Days | 1.3 (1.9) | 1.7 (2.0)
Statistical Analysis 1: Comparison: Drug-Coated Balloon (DCB) vs Standard PTA; Test type: Superiority or Other; p = 0.049, Chi-squared

ADVERSE EVENTS:
Arm/Group | Drug-Coated Balloon (DCB) | Standard PTA
Serious Adverse Events (participants affected / at risk) | 102/220 | 62/111
Other Adverse Events (participants affected / at risk) | 104/220 | 62/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-Coated Balloon (DCB) (N=220) | Standard PTA (N=111)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
MedDRA 13.0 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 2 (2) | 1 (1)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aorto-Duodenal Fistula (Vascular disorders) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (2) | 0 (0)
Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0)
Arterial Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Arterial Stenosis Limb (Vascular disorders) | 1 (1) | 3 (3)
Arterial Thrombosis Limb (Vascular disorders) | 0 (0) | 0 (0)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 2 (2)
Artery Dissection (Vascular disorders) | 7 (8) | 2 (2)
Arthritis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 6 (6) | 1 (1)
Carotid Artery Disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 7 (7) | 1 (1)
Coronary Artery Thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Device Occlusion (General disorders) | 1 (1) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0)
Diabetic Foot (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Diabetic Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Dry Gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolic Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Arterial Stenosis (Vascular disorders) | 15 (18) | 10 (12)
Femoral Artery Dissection (Vascular disorders) | 4 (4) | 5 (5)
Femoral Artery Occlusion (Vascular disorders) | 3 (5) | 5 (5)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured Coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Iliac Artery Occlusion (Vascular disorders) | 0 (0) | 0 (0)
Iliac Artery Stenosis (Vascular disorders) | 2 (2) | 1 (1)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 1 (2) | 1 (1)
Implant Site Thrombosis (General disorders) | 1 (1) | 0 (0)
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infected Lymphocele (Infections and infestations) | 1 (1) | 0 (0)
Intermittent Claudication (Vascular disorders) | 7 (7) | 11 (12)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0)
Multi-Organ Failure (General disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peptic Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 8 (8) | 5 (5)
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Peripheral Artery Dissection (Vascular disorders) | 3 (3) | 4 (5)
Peripheral Embolism (Vascular disorders) | 1 (1) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 2 (4) | 2 (2)
Peripheral Revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 2 (2) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic Specific Antigen Increased (Investigations) | 0 (0) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Subclavian Artery Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Therapeutic Embolisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 3 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vessel Puncture Site Haematoma (General disorders) | 2 (2) | 0 (0)
West Nile Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-Coated Balloon (DCB) (N=220) | Standard PTA (N=111)
Artery Dissection (Vascular disorders) | 46 (46) | 36 (37)
Femoral Artery Dissection (Vascular disorders) | 29 (29) | 11 (11)
Intermittent Claudication (Vascular disorders) | 0 (0) | 15 (16)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 21 (23) | 8 (8)
Peripheral Artery Dissection (Vascular disorders) | 14 (14) | 9 (11)
Vessel Puncture Site Haematoma (General disorders) | 13 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days